CLINICAL TRIAL: NCT03179631
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Efficacy and Safety Study of Ataluren in Patients With Nonsense Mutation Duchenne Muscular Dystrophy and Open-Label Extension
Brief Title: Long-Term Outcomes of Ataluren in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC124-GD-041-DMD
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Muscular Dystrophy, Duchenne; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Disease; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn
Keywords: Duchenne Muscular Dystrophy; Dystrophinopathy; Nonsense Mutation; Premature Stop Codon; Becker Muscular Dystrophy; DMD/BMD; PTC124; Ataluren
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn | interventions — ataluren

STUDY DESIGN:
Intervention Model Description: This study describes the randomized, double-blind, placebo-controlled, 72-week study and its 72-week open-label extension
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomized, double-blind, placebo-controlled,72-week study and its 72-week open-label extension
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ataluren (Experimental): 10, 20 milligrams per kilogram (mg/kg)
  Interventions: Drug: Ataluren
- Placebo (Placebo Comparator): 10, 20 mg/kg
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Ataluren — 10, 20 mg/kg
  Other Names: PTC124
  Arms: Ataluren
Drug: PLACEBO — 10, 20 mg/kg
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
This study is a long-term study of ataluren in participants with nonsense mutation Duchenne muscular dystrophy.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, 72-week study, followed by a 72-week open-label period. The purpose is to characterize the long-term effects of ataluren-mediated dystrophin restoration on disease progression. Participants will be randomized in a 1:1 ratio to ataluren or placebo. Participants will receive blinded study drug three times daily (TID) at morning, midday, and evening for 72 weeks, after which all participants will receive open-label ataluren for an additional 72 weeks (144 weeks in total). Study assessments will be performed at clinic visits every 12 weeks during the double-blind period and every 24 weeks during the open-label period. The total sample size of ~250 subjects will include ~160 subjects who meet the criteria for inclusion in the primary analysis population (age 7 to 16 years old, baseline six minute walk distance (6MWD) greater than or equal to (>=) 300 meters, supine to stand >= 5 seconds). The study will be conducted in the United States and other countries around the world.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age ≥5 years
* Phenotypic evidence of Duchenne Muscular Dystrophy
* Nonsense point mutation in the dystrophin gene
* Use of systemic corticosteroids (prednisone/prednisolone or deflazacort)for a minimum of 12 months immediately prior to start of study treatment, with no significant change in dosage or dosing regimen for a minimum of 3 months immediately prior to start of study treatment
* 6MWD ≥150 meters
* Ability to perform timed function tests within 30 seconds
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions.

Exclusion Criteria:

* Any change in prophylaxis treatment for cardiomyopathy within 1 month prior to start of study treatment.
* Ongoing intravenous (IV) aminoglycoside or IV vancomycin therapy.
* Prior or ongoing therapy with ataluren.
* Known hypersensitivity to any of the ingredients or excipients of the study drug
* Exposure to another investigational drug within 6 months prior to start of study treatment, or ongoing participation in any interventional clinical trial.
* History of major surgical procedure within 12 weeks prior to start of study treatment, or expectation of major surgical procedure during the 72-week placebo-controlled treatment period.
* Requirement for daytime ventilator assistance or any use of invasive mechanical ventilation via tracheostomy.
* Uncontrolled clinical symptoms and signs of congestive heart failure
* Elevated serum creatinine or cystatin C at screening.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Slope of Change in 6-Minute Walk Distance (6MWD) Over 72 Weeks | 72 weeks

SECONDARY OUTCOMES:
Change from Baseline to Week 72 in 6MWD | Baseline, Week 72
Change from Baseline to Week 72 in Time to Run/Walk 10 Meters | Baseline, Week 72
Change from Baseline to Week 72 in Time to Climb 4 Stairs | Baseline, Week 72
Change from Baseline to Week 72 in Time to Descend 4 Stairs | Baseline, Week 72
Change from Baseline to Week 72 in North Start Ambulatory Assessment (NSAA) Total Score | Baseline, Week 72
Time to Loss of Ambulation Over 72 Weeks | 72 weeks
Time to Loss of Stair-Climbing Over 72 Weeks | 72 Weeks
Time to Loss of Stair-Descending Over 72 Weeks | 72 weeks
Risk of Loss of NSAA Items Over 72 weeks | 72 weels
Number of Treatment-Emergent Adverse Events Considered Related to Study Drug | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Penematsa, MD, Study Director — PTC Therapeutics, Inc.
Locations (64):
- United States (22):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California, San Francisco (UCSF) - Benioff Children's Hospital - Oakland, Oakland, California
  - Stanford University Medical Center, Palo Alto, California
  - University of California (UC) Davis Medical Center, Sacramento, California
  - Loma Linda University Children's Hospital, San Bernardino, California
  - Northwest Florida Clinical Research Group, LLC, Gulf Breeze, Florida
  - Indiana University Health - Riley Child Neurology, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University College of Physicians & Surgeons, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriners Hospital for Children, Portland, Oregon
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Cook Childrens Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University Of Utah, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - The Childrens Hospital at Westmead, Westmead, New South Wales
  - The Royal Childrens Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
  - Queensland Children's Hospital, South Brisbane
- Brazil (3):
  - Hospital de Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo - FMUSP, São Paulo
- UMHAT Sofiamed, Sofia, Bulgaria
- Canada (2):
  - Childrens Hospital London Health Sciences Centre, London, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
- China (5):
  - General Hospital of Chinese Armed Police Forces, Beijing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Xiangya Hospital Central South University, Hunan
  - Children's Hospital of Fudan University, Shanghai
  - Shenzhen Children's Hospital, Shenzhen
- Queen Mary Hospital, Hong Kong, Hong Kong
- India (9):
  - Panchshil Hospital, Ahmedabad, Gujarat
  - National Institute of Mental Health and Neurosciences, Bengaluru, Karnataka
  - P.D. Hinduja Hospital, Māhīm, Maharashtra
  - Apollo Children's Hospital Chennai, Chennai, Tamil Nadu
  - Christian Medical College Hospital Vellore, Vellore, Tamil Nadu
  - Nizam's Institute of Medical Sciences (NIMS), Hyderabad, Telangana
  - Apollo Gleneagles Hospital, Kolkata, West Bengal
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - All India Institute of Medical Sciences, New Delhi
- PTC Clinical Site, Multiple Locations, Japan
- Malaysia (2):
  - Hospital Tunku Azizah Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre (UMMC), Pantai
- Mexico (3):
  - Hospital Angeles Chihuahua, Chihuahua City
  - Instituto Nacional de Pediatría, Mexico City
  - Instituto Nacional de Rehabilitacion, Tlalpan
- Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw, Poland
- University of Puerto Rico - School of Medicine, San Juan, Puerto Rico
- Russia (2):
  - Russian National Research Medical University n.a. N.I.Pirogov, structural branch - Research Clinical Institute of Pediatrics n.a. Academician Yu. E. Veltishchev, Moscow
  - "Saint Petersburg State Paediatric Medical University" based at Consultative and Diagnostic Centre, Saint Petersburg
- South Korea (3):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- Siriraj Hospital, Bangkok, Thailand
- Istanbul University- Instanbul Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: References — http://www.ptcbio.com